CLINICAL TRIAL: NCT00357565
Title: Hematopoietic Cell Transplantation in the Treatment of Infant Leukemia and Myelodysplastic Syndrome
Brief Title: Hematopoietic Stem Cell Transplantation in the Treatment of Infant Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005LS075; UMN-MT2005-25 (Other: Blood and Marrow Transplantation Program); UMN-0511M77206 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Childhood Acute Myeloid Leukemia in Remission; Recurrent Childhood Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Childhood Acute Lymphoblastic Leukemia in Remission; Previously Treated Myelodysplastic Syndrome; Secondary Myelodysplastic Syndrome; Refractory Anemia With Excess Blasts in Transformation; Refractory Anemia With Excess Blasts; Refractory Anemia; De Novo Myelodysplastic Syndrome; Childhood Myelodysplastic Syndrome
Keywords: MDS; AML
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Anemia, Refractory | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Busulfan; Cyclosporine; fludarabine phosphate; Melphalan; Mycophenolic Acid; Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Double Unit UCB Transplantation (Experimental): Patients that receive 2 units of umbilical cord blood transplantation (UCBT).
  Interventions: Biological: filgrastim; Drug: busulfan; Drug: cyclosporine; Drug: fludarabine phosphate; Drug: melphalan; Drug: mycophenolate mofetil; Procedure: umbilical cord blood transplantation
- Single Unit UCB Transplantation (Experimental): Patients that receive one unit of umbilical cord blood transplantation (only if 2 adequate size and matched units are not available).
  Interventions: Biological: filgrastim; Drug: busulfan; Drug: cyclosporine; Drug: fludarabine phosphate; Drug: melphalan; Drug: mycophenolate mofetil; Procedure: umbilical cord blood transplantation

INTERVENTIONS:
Biological: filgrastim — All patients will receive G-CSF 5 mcg/kg/day intravenous (IV) (dose rounded to vial size) based on the actual body weight IV beginning on day +1 after umbilical cord blood (UCB) infusion. G-CSF will be administered daily until the absolute neutrophil count (ANC) exceeds 2.5 x 10^9/L for three consecutive days and then discontinued. If the ANC decreases to <1.0 x 10^9/L, G-CSF will be reinstituted.
  Other Names: G-CSF
Drug: busulfan — Administered 1.1 mg/kg if <12 kg intravenous (IV) every 6 hours (0.8 mg/kg if >12 kg IV every 6 hours on Days -8 through -5.
  Other Names: Busulfex
Drug: cyclosporine — Patients will receive cyclosporine (CSA) therapy beginning on day -3 maintaining a level of >200 ng/mL. For children < 40 kg the initial dose will be 2.5 mg/kg intravenous (IV) over 2 hours every 8 hours.
  Other Names: CSA
Drug: fludarabine phosphate — Administered 25 mg/m^2 intravenous (IV) over 60 minutes on Days -4 through -2.
  Other Names: Fludara
Drug: melphalan — Administered 60 mg/m^2 intravenous (IV) over 30 minutes on Days -4 through -2.
  Other Names: Alkeran
Drug: mycophenolate mofetil — All patients will begin mycophenolate mofetil (MMF) on day -3. Patients <45 kilograms will receive MMF at the dose of 15 mg/kg/dose every 8 hours (max dose 1gm/dose) orally or intravenously (PO or IV).
  Other Names: MMF
Procedure: umbilical cord blood transplantation — The product is infused via IV drip directly into the central line without a needle, pump or filter on Day 0.

SUMMARY:
RATIONALE: Giving chemotherapy, such as busulfan, fludarabine, and melphalan, before a donor umbilical cord blood stem cell transplant helps stop the growth of abnormal or cancer cells and prepares the patient's bone marrow for the stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil may stop this from happening.

PURPOSE: This phase II trial is studying how well combination chemotherapy followed by a donor umbilical cord blood transplant works in treating infants with high-risk acute leukemia or myelodysplastic syndromes.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the incidence of engraftment, defined as achieving donor-derived neutrophil count > 500/mm³ by day 42, in infants with high-risk acute myeloid leukemia, acute lymphoblastic leukemia, or myelodysplastic syndromes treated with a non-irradiation containing myeloablative conditioning regimen comprising busulfan, fludarabine, and melphalan followed by double umbilical cord blood transplantation (UCBT) with two partially HLA-matched units.

Secondary Objectives

* Determine the incidence of transplant-related mortality (TRM) at 6 months after UCBT
* Evaluate pattern of chimerism after double UCBT
* Determine the incidence of platelet engraftment at 1 year after UCBT
* Determine the incidence of acute graft-versus-host disease (GVHD) grade II-IV and grade III-IV at day 100 after UCBT
* Evaluate the developmental outcome after UCBT

Transplant Related Objectives

* Determine the incidence of chronic GVHD at 1 year after UCBT
* Determine the survival and disease free survival at 1 and 2 years after UCBT
* Determine the incidence relapse at 1 and 2 years after UCBT

ELIGIBILITY:
Inclusion Criteria:

* Matched sibling donor (HLA 8/8), if available, or a unrelated partially HLA matched single unit based on the following priority:

  * 1st priority: 4/6 matched unit, cell dose >5 x 10-7 nucleated cells/kg
  * 2nd priority: 5/6 matched unit, cell dose > 4 x 10-7 nucleated cells/kg
  * 3rd priority: 6/6 matched unit, cell dose > 3 x 10-7 nucleated cells/kg
* Patients aged ≤ 3 years at diagnosis (not age of transplant) with hematological malignancy as detailed below:

  * Acute myeloid leukemia: high risk CR1 as evidenced by:

    * High risk cytogenetics t(4;11) or other MLL rearrangements; chromosome 5, 7, or 19 abnormalities; complex karyotype (>5 distinct changes); ≥ 2 cycles to obtain complete response (CR); CR2 or higher; Preceding myelodysplastic syndrome (MDS); All patients must be in CR or early relapse (i.e., <15% blasts in BM).
    * Acute lymphocytic leukemia: high risk CR1 as evidenced by: High-risk cytogenetic: t(4;11) or other MLL rearrangements; hypodiploid; t(9;22); >1 cycle to obtain CR; CR2 or higher; All patients must be in CR as defined by hematological recovery, AND <5% blasts by light microscopy within the bone marrow with a cellularity of ≥15%.
  * Myelodysplasia (MDS) IPSS Int-2 or High risk (i.e. RAEB, RAEBt) or refractory anemia with severe pancytopenia or high risk cytogenetics. Blasts must be < 10% by a representative bone marrow aspirate morphology.
  * Persistent or rising minimal residual disease (MRD) after standard chemotherapy regimens: Patients with evidence of minimal residual disease at the completion of therapy or evidence of rising MRD while on therapy. MRD will be defined by either flow cytometry (>0.1% residual cells in the blast gate with immune phenotype of original leukemic clone), by molecular techniques (PCR or FISH) or conventional cytogenetics (g-banding).
  * New Leukemia Subtypes: A major effort in the field of pediatric hematology is to identify patients who are of high risk for treatment failure so that patients can be appropriately stratified to either more (or less) intensive therapy. This effort is continually ongoing and retrospective studies identify new disease features or characteristics that are associated with treatment outcomes. Therefore, if new high risk features are identified after the writing of this protocol, patients can be enrolled with the approval of two members of the study committee.
* Recipients must have a Lansky score ≥ 50% and have acceptable organ function defined as:

  * Renal: glomerial filtration rate > 60ml/min/1.73m^2
  * Hepatic: bilirubin, AST/ALT, ALP < 5 x upper limit of normal,
  * Pulmonary function: oxygen saturation >92%
  * Cardiac: left ventricular ejection fraction > 45%.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care.

Exclusion Criteria:

* Active infection at time of transplantation (including active infection with Aspergillus or other mold within 30 days).
* History of HIV infection or known positive serology
* Myeloablative transplant within the last 6 months.
* Evidence of active extramedullary disease (including central nervous system leukemia).

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2005-11 (Actual); Primary Completion 2024-06 (Actual); Study Completion 2025-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christen Ebens, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- BM Transplantation: Blood and Marrow transplantation
Period: Overall Study
Arm/Group | Double Unit UCB Transplantation | Single Unit UCB Transplantation | BM Transplantation
Started | 15 | 15 | 4
Completed | 15 | 15 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double Unit UCB Transplantation | Single Unit UCB Transplantation | BM Transplantation | Total
Number analyzed (Participants) | 15 | 15 | 4 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 15 | 4 | 34
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 4 | 17
  Male | 7 | 10 | 0 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 12 | 14 | 4 | 30
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 2 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 10 | 13 | 3 | 26
  More than one race | 2 | 0 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 4 | 34

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Engraftment
Description: Defined as achieving donor derived neutrophil count >500/uL by day 42 in young children with leukemia or myelodysplastic syndrome undergoing a partially matched single unit umbilical cord blood transplant (UCBT) after a myeloablative preparative regimen consisting of busulfan, melphalan and fludarabine.
Time Frame: Day 42 After Transplant
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Double Unit UCB Transplantation | Single Unit UCB Transplantation | BM Transplantation
Number analyzed (Participants) | 15 | 15 | 4
Percentage of participants | 100 [0 to 100] | 93 [42 to 99] | 100 [0 to 100]

2. Secondary Outcome: Incidence of Transplant-related Mortality (TRM)
Description: defined as death due to transplant
Time Frame: at 6 months after transplant
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Double Unit UCB Transplantation | Single Unit UCB Transplantation | BM Transplantation
Number analyzed (Participants) | 15 | 15 | 4
Percentage of participants | 33 [11 to 57] | 13 [2 to 35] | 0 [0 to 0]

3. Secondary Outcome: Incidence of Platelet Engraftment
Description: defined as platelet count > 50,000
Time Frame: at 1 year after transplant
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Double Unit UCB Transplantation | Single Unit UCB Transplantation | BM Transplantation
Number analyzed (Participants) | 15 | 15 | 4
Percentage of participants | 80 [8 to 98] | 100 [0 to 100] | 100 [0 to 100]

4. Secondary Outcome: Incidence of Acute Graft-versus-host Disease (GVHD) Grade II-IV and Grade III-IV
Description: Graft-versus-host disease (GVHD) is a common complication of allogeneic bone marrow transplantation in which functional immune cells in the transplanted marrow recognize the recipient as "foreign" and mount an immunologic attack.
Time Frame: Day 100 After Transplant
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Double Unit UCB Transplantation | Single Unit UCB Transplantation | BM Transplantation
Number analyzed (Participants) | 15 | 15 | 4
Percentage of participants | 40 [16 to 64] | 33 [11 to 57] | 0 [0 to 0]

5. Secondary Outcome: Incidence of Chronic Graft-versus-host Disease (GVHD)
Description: as for outcome 4
Time Frame: 1 Year After Transplant
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Double Unit UCB Transplantation | Single Unit UCB Transplantation | BM Transplantation
Number analyzed (Participants) | 15 | 15 | 4
Percentage of participants | 13 [1 to 40] | 0 [0 to 0] | 0 [0 to 0]

6. Secondary Outcome: Incidence of Relapse
Description: defined using standard criteria (bone marrow blast count and cytogenetics).
Time Frame: 1 and 2 years after transplant
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Double Unit UCB Transplantation | Single Unit UCB Transplantation | BM Transplantation
Number analyzed (Participants) | 15 | 15 | 4
Percentage of participants
  1 year | 13 [2 to 35] | 20 [4 to 43] | 0 [0 to 0]
  2 years | 13 [2 to 35] | 20 [4 to 43] | 25 [0 to 83]

7. Secondary Outcome: Overall Survival
Description: Alive after transplant.
Time Frame: at 1 and 2 years after transplant
Measure: Number (95% Confidence Interval); unit: Probability of survival
Arm/Group | Double Unit UCB Transplantation | Single Unit UCB Transplantation | BM Transplantation
Number analyzed (Participants) | 15 | 15 | 4
Probability of survival
  1 year | 0.53 [0.33 to 0.86] | 0.67 [0.47 to 0.95] | 100 [100 to 100]
  2 years | 0.47 [0.27 to 0.80] | 0.67 [0.47 to 0.95] | 0.67 [0.3 to 1]

8. Secondary Outcome: Disease-free Survival
Description: defined as patients who are alive and in hematological remission.
Time Frame: at 1 and 2 years after transplant
Measure: Number (95% Confidence Interval); unit: Probability of survival
Arm/Group | Double Unit UCB Transplantation | Single Unit UCB Transplantation | BM Transplantation
Number analyzed (Participants) | 15 | 15 | 4
Probability of survival
  1 year | 0.13 [0.02 to 0.35] | 0.2 [0.04 to 0.43] | 0 [0 to 0]
  2 years | 0.13 [0.02 to 0.35] | 0.20 [0.04 to 0.43] | 0.33 [0 to 0.83]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Double Unit UCB Transplantation | Single Unit UCB Transplantation | BM Transplantation
All-Cause Mortality (participants affected / at risk) | 8/15 | 5/15 | 1/4
Serious Adverse Events (participants affected / at risk) | 8/15 | 5/15 | 1/4
Other Adverse Events (participants affected / at risk) | 15/15 | 15/15 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Unit UCB Transplantation (N=15) | Single Unit UCB Transplantation (N=15) | BM Transplantation (N=4)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Leukemia relapse (Investigations) | 2 (2) | 3 (3) | 1 (1)
Respiratory failure (any cause) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Multi-organ Failure (Investigations) | 2 (2) | 1 (1) | 0 (0)
Chronic Graft versus host disease (Investigations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Unit UCB Transplantation (N=15) | Single Unit UCB Transplantation (N=15) | BM Transplantation (N=4)
PERICARDIAL EFFUSION (Cardiac disorders) | 4 (4) | 2 (2) | 0 (0)
Renal replacement therapy / dialysis (Renal and urinary disorders) | 3 (4) | 3 (3) | 0 (0)
Veno-Occlusive Disease (Hepatobiliary disorders) | 4 (4) | 5 (6) | 0 (0)
Respiratory failure requiring intubation/ventilation (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4) | 0 (0)
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Viremia (Infections and infestations) | 6 (6) | 2 (2) | 2 (2)
Gram positive bacteremia (Infections and infestations) | 6 (6) | 3 (3) | 1 (1)
Gram negative bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Pneumonia (Infections and infestations) | 7 (7) | 5 (5) | 0 (0)
Graft versus host disease grade 1-2 (Investigations) | 2 (2) | 3 (3) | 1 (1)
Chronic Graft versus host disease (Investigations) | 2 (2) | 0 (0) | 0 (0)
Graft versus host disease grade 3-4 (Investigations) | 4 (4) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/65/NCT00357565/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/65/NCT00357565/ICF_001.pdf